CLINICAL TRIAL: NCT03628625
Title: Letrozole Pretreatment With Misoprostol for Induction of Abortion In First-Trimester Missed Miscarriage: A Randomized Controlled Trial
Brief Title: Letrozole Pretreatment With Misoprostol fInduction of Abortion In First-Trimester Missed Miscarriage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr- dina yahia mansour, Lecturer of Obstetrics and Gynecology Ain Shams University, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0005
Record Dates: First submitted 2018-05-10; First posted 2018-08-14 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Miscarriage; Missed Abortion
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed | interventions — Letrozole; Misoprostol

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): 3 tablets of Letrozole 2.5 mg will be given as single daily dose, 7.5 mg per day for two days at home and the third dose will be given on admission to hospital on day 3 and will be followed by vaginal misoprostol 800 mcg every three hours up to maximum two doses.
  Interventions: Drug: Letrozole 2.5mg; Drug: Misoprostol
- Control group (Placebo Comparator): three tablets of placebo will be given as a single daily dose, for two days at home and will be admitted on day 3 and continue treatment with misoprostol 800 mcg every three hours up to maximum two doses
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Letrozole 2.5mg — total dose 7.5 mg per day for 3 days
  Arms: Study group
Drug: Placebo — Folic acid for 3 days
  Arms: Control group
Drug: Misoprostol — Misoprosrol 800mcg will be given to all patients for induction of abortion

SUMMARY:
This study compares the success rate of letrozole and misoprostol versus misoprostol alone for medical termination of first trimester pregnancy.

DETAILED DESCRIPTION:
According to the American college of obstetricians and gynecologists (2005), medical abortion is an acceptable alternative for surgical procedures in pregnant women with gestational age of less than 49 days based on the last menstrual period

Oral or vaginal misoprostol causes complete abortion in almost 85% of cases within seven days before the 12th week

letrozole administration with misoprostol raises the rate of complete abortion

Hypothesis:

In women with missed miscarriage in the first trimester undergoing induction of abortion pre-treatment with letrozole before misoprostol may lead to abortion rate similar to misoprostol alone.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 64 days gestation (<9 wks).
* Hemoglobin >10 g/dL.
* BMI between 18.5 kg/m2 and 25 kg/m2.
* Missed abortion.

Exclusion Criteria:

* Molar pregnancy.
* Fibroid uterus.
* Uterine anomalies.
* Coagulopathy.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-12-05 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete miscarriage | 6 hours

SECONDARY OUTCOMES:
Need for surgical evacuation of the products of conception | 6 hours
Incidence of Septic Abortion | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Egypt